CLINICAL TRIAL: NCT05136378
Title: Administration of Selenious Yeast Tablets in Chronic Lymphocytic Leukemia Patients Without Indication of Chemotherapy: A Multicenter Study
Brief Title: Selenious Yeast in CLL Patients w/o Indication of Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020ZSLC56; B2021-447R (Other: EC, Zhongshan Hospital)
Record Dates: First submitted 2021-11-23; First posted 2021-11-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Chronic Lymphocytic Leukemia Stage A(0); Chronic Lymphocytic Leukemia Stage A(I); Chronic Lymphocytic Leukemia Stage A(II); Chronic Lymphocytic Leukaemia Stage B(I)
Keywords: Chronic Lymphocytic Leukemia; Humans; Prospective Studies; Selenium
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (No Intervention): Wait and Watch.
- Low Dose Selenious Yeast (Experimental): Receive 200μg Selenious Yeast per day.
  Interventions: Drug: Low Dose Selenious Yeast Tablets
- High Dose Selenious Yeast (Experimental): Receive 400μg Selenious Yeast per day.
  Interventions: Drug: High Dose Selenious Yeast Tablets

INTERVENTIONS:
Drug: Low Dose Selenious Yeast Tablets — Low dose of Selenious Yeast Tablets
  Arms: Low Dose Selenious Yeast
Drug: High Dose Selenious Yeast Tablets — High Dose Selenious Yeast Tablets
  Arms: High Dose Selenious Yeast

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Selenious Yeast Tablets in Chronic Lymphocytic Leukemia Patients without Indication of Chemotherapy

DETAILED DESCRIPTION:
A large portion of CLL patients has no indications of chemotherapy when diagnosed. In patients with CLL, the mean serum selenium levels are lower than normal. There is a correlation between the selenium level and the clinical stage. We discovered that sodium selenite inhibited the expression of CXCL-1 and restored the defective necroptotic pathway of CLL cells together with TNF-α and z-VAD in vitro. The purpose of this study is to evaluate the safety and effectiveness of Selenious Yeast Tablets in preventing CLL patients without indication of chemotherapy from disease development.

ELIGIBILITY:
Inclusion Criteria:

-

Newly diagnosed CLL/small lymphocytic lymphoma (SLL) that meets criteria below:

1. Newly diagnosed (< 12 months from pre-registration on this study) CLL according to the National Cancer Institute (NCI) criteria or SLL according to the World Health Organization (WHO) criteria; this includes previous documentation of: Biopsy-proven small lymphocytic lymphoma OR Diagnosis of CLL according to NCI working group criteria as evidenced by all of the following: Peripheral blood lymphocyte count of > 5,000/mm^3; if present, prolymphocytes should be < 55% AND Immunophenotyping consistent with CLL defined as:The predominant population of lymphocytes share both B-cell antigens (cluster of differentiation [CD]19, CD20, or CD23) as well as CD5 in the absence of other pan-T-cell markers (CD3, CD2, etc.) Dim surface immunoglobulin expression Restricted surface kappa or lambda light chain expression Before diagnosing CLL or SLL, mantle cell lymphoma must be excluded by demonstrating a negative fluorescent in situ hybridization (FISH) analysis for t(11;14)(immunoglobulin H [IgH]/cyclin D 1 [CCND1]) on peripheral blood or tissue biopsy or negative immunohistochemical stains for cyclin D1 on involved tissue biopsy
2. Rai stage 0 or 1
3. Previously untreated
4. Asymptomatic with the plan for observation(NOT meet iwCLL indication of chemotherapy)
5. Life expectancy of at least 12 months
6. Willing to provide tissue for correlative research purpose

Exclusion Criteria:

1. Concentration of serum Se exceed the normal range
2. Active other malignancy requiring treatment that would interfere with the assessments of this study
3. Hepatitis B or C
4. Autoimmune disease history
5. Organ transplant recipients need to receive drug therapy
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 17 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year DPR | 2 years from enrollment
  2-year Disease Progression Rate
Decrease rate of Lymphocyte | 2 years from enrollment
  Decrease rate of peripheral lymphocyte counts

SECONDARY OUTCOMES:
Selenium Concentration, Serum | Enrollment, 1 Month(from enrollment), 3 Months, 6 Months
  Serum selenium concentration
adverse events | Enrollment, 1 Month (from enrollment), 3 Months, 6 Months
  safety profile of the subjects from enrollment
progression free survival (PFS) | 2 years from enrollment
overall survival (OS) | 2 years from enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China